CLINICAL TRIAL: NCT05890950
Title: A 28-Day Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of K-757 and K-833 in Overweight/Obese Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of K-757 and K-833 in Overweight/Obese Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kallyope Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K-757 P005
Record Dates: First submitted 2023-04-07; First posted 2023-06-06 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Obesity; Type 2 Diabetes Mellitus in Obese
Keywords: Obesity; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- K-757 and K-833 combination (Experimental)
  Interventions: Drug: K-757 and K-833
- Placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo to K-757 and K-833

INTERVENTIONS:
Drug: K-757 and K-833 — Both administered orally
  Arms: K-757 and K-833 combination
Drug: Matching placebo to K-757 and K-833 — Both administered orally
  Arms: Placebo

SUMMARY:
This is a multiple dose study to evaluate the safety, tolerability, PK, and PD of K-757 and K-833 when co-administered in overweight/obese patients with Type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

1. Understand the trial procedures and agree to participate by providing written informed consent.
2. Be willing and able to comply with all trial procedures and restrictions, including following study diet requirements.
3. Be between 18 to 70 years of age, inclusive, at the Screening Visit.
4. Has T2DM in accordance with American Diabetes Association (ADA) guidelines at Screening.
5. Is on stable metformin monotherapy (total daily dose of 500 to 2,000 mg/day) for at least 3 months and tolerating metformin well in the opinion of the investigator. Note: Both the immediate release (IR) and extended release (XR) formulations of metformin are acceptable.
6. HbA1c of 7.0% to 10.5% at Screening.
7. Have a Body Mass Index (BMI) ≥25.0 and <38.0 (kg/m2) at the Screening Visit.
8. Be weight stable (<5% variation) over the last 3 months, by subject report.
9. Be a nonsmoker who has not used tobacco or nicotine-containing products (e.g. nicotine patch, e-cigarettes, vapes) for at least 3 months before administration of the initial dose of trial drug and agrees to abstain from smoking tobacco or the use of nicotine-containing products while on study.
10. Be judged to be in generally good health by the Investigator, based on clinical evaluations including laboratory safety tests, medical history, physical examination, 12-lead ECG, and vital sign measurements performed at the Screening Visit and before administration of the initial dose of trial drug.
11. Meet the following requirements:

    1. Is a male who agrees to all of the following:

       * To use an appropriate method of contraception, including a condom with or without spermicidal cream or jelly, from the first dose of study drug until 14 days after the last dose of study drug. A male subject who had a vasectomy procedure must follow the same restrictions as a non-vasectomized man.
       * If partner is pregnant, to use a condom.
       * To not donate sperm from the first dose of study drug until 14 days after the last dose of study drug.

       OR
    2. Is a female who is of non-childbearing potential defined by at least 1 of the following criteria:

       * Postmenopausal (aged >45 years and with a minimum of 12 months of spontaneous amenorrhea with a Screening serum follicle-stimulating hormone (FSH) level in the menopausal range as established for the laboratory performing the test.
       * Post hysterectomy, bilateral oophorectomy or bilateral salpingectomy, based on the subject's recall of their medical history.

       OR
    3. Is a female of reproductive potential and:

       * agrees to remain abstinent from heterosexual activity or
       * agrees to use (or have their partner use) a birth control method that is highly effective and has low user dependency. Acceptable methods of birth control are:

         * Progestogen-only implant (e.g. etonogestrel implant)
         * Intrauterine device (IUD)
         * Intrauterine hormone-releasing system (IUS)
         * Bilateral tubal occlusion
         * Vasectomized partner

Exclusion Criteria:

1. Has participated in another interventional investigational study within 30 days of the Screening Visit. The window will be derived from the date of the last study procedure and/or AE related to the study procedure in the previous study to the Screening Visit of the current study. If the subject received an investigational medication in the prior study, at least 5 half-lives (or longer if required by local regulations) must have passed between the last dose of the investigational product and the Screening Visit.
2. Is an employee or immediate family member (eg, spouse, parent, child, sibling) of the Sponsor or study site.
3. Has a history of multiple significant and/or any severe allergies (eg, food, drug, latex allergy) or has had an anaphylactic reaction or significant intolerance to prescription or nonprescription drugs or food.
4. Has a known hypersensitivity or contraindication to any component of K-757 or K-833, including excipients.
5. Has a positive alcohol or drug screen at Screening or admission.
6. Has a positive pregnancy test.
7. Is a lactating/nursing female.
8. Has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency antibody, at the Screening Visit. Note: Subjects with positive hepatitis B virus or hepatitis C virus serology may be enrolled if quantitative polymerase chain reaction for hepatitis B virus or hepatitis C virus ribonucleic acid is negative.
9. Does not meet study site COVID-19 admission/study participation restrictions.
10. Has a fever (>38oC).*
11. Had major surgery or donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the Screening Visit.*
12. Is unable to refrain from the use of prohibited prescription or non-prescription drugs including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication through completion of study participation.

    As detailed in Section 10.1, allowable concomitant medications may include HMG-CoA reductase inhibitors (statins), ≤2 permissible anti-hypertensive agents, postmenopausal hormone replacement therapy, and/or proton pump inhibitors (PPIs).
13. Has been on any GLP-1 receptor agonist, any dipeptidyl peptidase IV (DPP-4) inhibitor, or any approved or investigational medications known to cause weight loss in the prior 3 months.
14. Has a history of type 1 diabetes mellitus (T1DM) or a history of diabetic ketoacidosis or subject assessed by the investigator as possibly having T1DM.
15. Has a history of other specific types of other specific types of diabetes (e.g. genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrinopathies, drug- or chemical-induced, and post organ transplant diabetes).
16. Has been treated with insulin or any other AHAs other than metformin within 4 weeks of screening or within 12 weeks of screening if the AHA was a thiazolidinedione (e.g., rosiglitazone, pioglitazone).
17. At Screening or Day -1 has a site fasting fingerstick glucose of >270 mg/dL.*
18. Has evidence or history of diabetic complications or significant end organ damage, eg, proliferative retinopathy and/or macular edema, eGFR (MDRD) ≤60 mL/min, diabetic neuropathy.
19. One or more self-reported episodes of hypoglycemia (fingerstick glucose <60 mg/dL with symptoms consistent with hypoglycemia or <50 mg/dL irrespective of symptoms) within the last 3 months.
20. Is using or anticipates the need for using concomitant medications which are inhibitors of P-gp or BCRP or any prohibited medications from screening until the post study visit.
21. Has excessive consumption of alcohol within 6 months prior to screening (>14 drinks/week for men and >7 drinks/week for women, where l drink= 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) or use any of soft drugs(such as marijuana) within 3 months prior to Screening, or hard drugs (such as cocaine) within 6 months prior to Screening.
22. Is unwilling or unable to refrain from consuming alcohol from 7 days prior to the first dose of study medication through the completion of study participation.
23. Has a substance abuse disorder.
24. Had a previous major psychotic disorder.
25. Has a corrected QT interval to Fridericia's formula (QTcF) >450 milliseconds (msec) for males and >470 msec for females at screening or admission.
26. Has a mean value for triplicate semi-recumbent systolic blood pressure >160 millimeters of mercury (mmHg) and/or diastolic blood pressure (BP) >95 mmHg measured after at least 10 minutes at rest at the Screening Visit. Note: If a subject's BP is exclusionary on the first triplicate assessment at the Screening visit, they may have 1 repeat triplicate BP assessment at that visit, after another rest of at least 10 minutes, to qualify for the study.

    If a subject's BP is exclusionary at screening but the investigator feels that BP is likely to be below the exclusionary thresholds at admission (Day -2), this criterion can be re-assessed at admission. Adjustment of doses of anti-hypertensives already being taken at screening is permissible, but initiation of new agents is not permissible. For subjects whose BP is exclusionary at Screening and at the first triplicate assessment on Day -2, triplicate assessments can be repeated up to twice on Day -2, as needed.
27. Has alanine aminotransferase or aspartate aminotransferase (ALT or AST) of >1.0X upper limit of normal (ULN) or total bilirubin >1.2X ULN (isolated bilirubin >1.2X ULN is acceptable if bilirubin is fractionated, and direct bilirubin is within the laboratory normal range) at Screening or admission. (Note: Subjects who do not meet this criterion at Screening or at admission may not be rescreened/retested).
28. Has serum amylase or lipase >1.2X the ULN at the Screening Visit.
29. Has a recent history (within past 3 years) or current diagnosis of any of the following GI (gastro-intestinal) related diseases: intestinal obstruction, GI perforation, GI motility disorders, adhesions, Clostridium difficile colitis or have had recent unexplained GI bleeding within 3 months prior to screening.
30. Has any history of pancreatitis (acute or chronic), gastroparesis, ischemic colitis, inflammatory bowel disease (IBD), celiac disease, irritable bowel syndrome (IBS), or colitis.
31. Has any past surgical history of gastric banding or bariatric surgery or bowel resection.
32. Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, neurologic disorder, neoplastic, or genitourinary abnormalities or diseases.
33. Has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the subject by their participation in the study.

note - *Subject may be included if they are able to return to the site within 7 days of initial screening and the exclusion criterion is no longer met.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who experienced 1 or more treatment-emergent AEs | Up to Day 42 +/- 2days
  After treatment with the combination of K-757 and K-833
Proportion of participants who discontinued study medication due to an AE | Up to Day 42 +/- 2days
  After treatment with the combination of K-757 and K-833

SECONDARY OUTCOMES:
Area under the concentration-time curve [AUC] of plasma K-757 | Days 14 and 28
  when co-administered with K-833
AUC of plasma K-833 | Days 14 and 28
  when co-administered with K-757
Maximum concentration [Cmax] of plasma K-757 | Days 14 and 28
  when co-administered with K-833
Cmax of plasma K-833 | Days 14 and 28
  when co-administered with K-757
Time of maximum concentration [Tmax] of plasma K-757 | Days 14 and 28
  when co-administered with K-833
Tmax of plasma K-833 | Days 14 and 28
  when co-administered with K-757
Clearance [Cl] of plasma K-757 | Days 14 and 28
  when co-administered with K-833
Cl of plasma K-833 | Days 14 and 28
  when co-administered with K-757
Volume of distribution at steady-state [Vdss] of plasma K-757 | Days 14 and 28
  when co-administered with K-833
Vdss of plasma K-833 | Days 14 and 28
  when co-administered with K-757
Half-life [t1/2] of plasma K-757 | Days 14 and 28
  when co-administered with K-833
t1/2 of plasma K-833 | Days 14 and 28
  when co-administered with K-757

CONTACTS AND LOCATIONS:
Locations (1):
- QPS, LLC, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No